CLINICAL TRIAL: NCT01765153
Title: Precision Versus Endurance Training to Improve Walking After Chronic Incomplete SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00003873
Record Dates: First submitted 2012-11-30; First posted 2013-01-10 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-01

CONDITIONS: Spinal Cord Injury
Keywords: physical therapy; rehabilitation; neuroplasticity
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endurance first (Experimental): Participants to start with Endurance Training. Participants are trained daily to walk on a treadmill for as fast and as long as possible. A harness supporting part of their body weight can be used if needed. Assistance from a trainer is used if needed. A physical therapist supervises the training. Training was 5x/wk for 2 months, followed by a 2-month rest period. Participants then returned for training in the Precision Training 5x/wk for 2 months.Participants train to walk over ground on 15 m straight hallway with obstacles they must step over, and targets they must step onto. This is followed by another 2-month rest. Measures of walking speed, distance, skill, confidence, as well as mood were obtained at least 3 times before any training, then monthly thereafter.
  Interventions: Behavioral: Endurance; Behavioral: Precision
- Precision first (Experimental): Participants to start with Precision Training. Participants train to walk over ground on 15 m straight hallway with obstacles they must step over, and targets they must step onto. Training was 5x/wk for 2 months, followed by a 2-month rest period. Participants then returned for Endurance Training 5x/wk for 2 months. Participants are trained to walk on a treadmill for as fast and as long as possible. A harness supporting part of their body weight can be used if needed. Assistance from a trainer is used if needed. A physical therapist supervises the training. followed by another 2-month rest. Measures of walking speed, distance, skill, confidence, as well as mood were obtained at least 3 times before any training, then monthly thereafter.
  Interventions: Behavioral: Endurance; Behavioral: Precision

INTERVENTIONS:
Behavioral: Endurance — Participants are trained daily to walk on a treadmill for as fast and as long as possible. A harness supporting part of their body weight can be used if needed. Assistance from a trainer is used if needed. A physical therapist supervises the training.
  Other Names: Treadmill walking training; Body-weight supported treadmill training
Behavioral: Precision — Participants train daily to walk over ground on 15 m straight hallway with obstacles they must step over, and targets they must step onto.
  Other Names: Skill walking training

SUMMARY:
The objective of the study was to determine the efficacy of two forms of physical therapy training, one emphasizing precise, visually guided walking over obstacles and on targets (Precision Training), the other emphasizing mass practice of walking on a treadmill (Endurance Training). The hypothesis was that visually guided training (Precision) may be especially efficacious because it engages the motor cortex, whose input may facilitate improvements in functional walking. Participants are individuals with a chronic (≥7 months post-injury), motor incomplete spinal cord injury (SCI), with no other problems that would preclude participation in an intensive training program. A randomized, single-blinded, cross-over design was used to randomly allocate participants to start with Precision or Endurance Training, identified as Training Phase I. Training was 5x/wk for 2 months, followed by a 2-month rest period, identified as Rest Period I. Participants then returned for 2-months of training in the other method, identified as Training Phase II, followed by another 2-month rest, Rest Period II. Measures of walking speed, distance, skill, confidence, as well as depression were obtained at least 3 times before any training, then monthly thereafter. Electrophysiological measures were taken before and after each phase of training and period of rest. Change scores were used to determine how each phase of training and rest influenced the scores (see below).

DETAILED DESCRIPTION:
PARTICIPANTS: Inclusion criteria: 1) SCI from trauma or other stable lesions, 2) injury occurred ≥ 7 mo prior, 3) able to walk independently at least 5 m with a walking aid and/or braces, 4) injury level between C1-L1, 5) able to give informed consent, 6) able to attend training sessions 5x/week. Exclusion criteria: 1) head injury, 2) cognitive or musculoskeletal impairments that preclude participation in walking training, 3) seizures or implants in the head that would preclude participation in experiments using transcranial magnetic stimulation (TMS).

INTERVENTIONS:

Precision Training. Training was performed on a 15 m long track. The track contained obstacles and targets. Obstacles were made of Styrofoam blocks of 3 cm height each, varying in width from 4 cm to 20 cm in divisions of 4 cm increments (which must be cleared without touching), and targets were made of fabric circles, ranging in diameter from 7-10.5 cm (which must be totally obscured by their foot). The difficulty of the track was designed to have the participant achieve ~80% success. The emphasis was on accuracy, not speed.

Endurance Training. The aim of this training was mass practice. Participants walked on the treadmill, with body-weight support (BWS) and manual assistance if needed. The treadmill speed was initially set to be faster than their over ground walking speed as measured by the 10 MWT(ss). Participants were encouraged to walk for as far and as fast as possible with minimal rest periods. Progression involved reducing manual assistance and BWS, increasing walking speed and distance, while reducing rest breaks.

In both phases of training, a research assistant or volunteer recorded training parameters each session. The number of steps executed was measured with a step counter (StepWatch, Orthocare Innovations, USA), which was confirmed to be accurate with simultaneous manual counting prior to its use, and periodically during training sessions. The heart rate before and immediately after each bout of walking was measured with a heart rate monitor (Polar FT7, Polar, Canada). The total time, distance and walking speed for each walking bout was recorded.

MEASURES:

Measures were taken prior to all training at baseline (called Baseline I) and the end of each of the following intervals - one month of Training Phase I, two months of Training Phase I, one month of Rest Period I, two months of Rest Period I, one month of Training Phase II, two months of Training Phase II, one month of Rest Period II, two months of Rest Period II. To measure changes during the second phase of training, the baseline was the average of the one and two month measures of Rest Period I, henceforth called Baseline II.

STATISTICAL ANALYSIS: To determined if one type of training was superior to the other, we compared the change scores (i.e., post-training score minus pre-training score) from each type of training using a standard t-test or a Mann-Whitney U test, as appropriate. Since individuals with high compared to low walking function may respond to the training differently, we divided individuals based on their pretraining walking speed as measured by the 10 MWT(ss) (i.e., > or < 0.5 m/s). The change scores from each of these groups of individuals were then compared for each type of training using a standard t-test or a Mann-Whitney U test, as appropriate. To determine the time course for obtaining a treatment effect, we compared the change scores for the first month (i.e., outcome measure at end of 1 mo minus baseline) versus the second month (outcome measure at end of 2 mo minus at end of 1 mo) of training for each type of training, using a standard t-test or a Mann-Whitney U test, as appropriate. Retention of gains was followed for 2 months after each type of training. The outcome measures at the end of the 2 month rest period were compared to the measures immediately after the training, for individuals that made improvements greater than the standard error of measurement for each measure, using a paired t-test or Wilcoxon signed-rank test, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* spinal cord injury equal or more than 7 months prior
* able to walk at least 5 meters independently (can use walking aids and braces)
* injury level between C1 and L1
* able to give informed consent
* able to attend training sessions 5x/week

Exclusion Criteria:

* head injury
* cognitive of musculoskeletal impairments that preclude participation in walking training
* seizures or implants in the head that would preclude participation in experiments with transcranial magnetic stimulation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaynie Yang, PhD, Principal Investigator — University of Alberta; Monica Gorassini, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Khan AS, Patrick SK, Roy FD, Gorassini MA, Yang JF. Training-Specific Neural Plasticity in Spinal Reflexes after Incomplete Spinal Cord Injury. Neural Plast. 2016;2016:6718763. doi: 10.1155/2016/6718763. Epub 2016 Sep 20. PMID 27725887
- [Derived] Musselman KE, Yang JF. Spinal Cord Injury Functional Ambulation Profile: a preliminary look at responsiveness. Phys Ther. 2014 Feb;94(2):240-50. doi: 10.2522/ptj.20130071. Epub 2013 Oct 10. PMID 24114437

RESULTS

PARTICIPANT FLOW:
Groups:
- Endurance First: Participants start with Endurance Training. Participants trained daily to walk on a treadmill for as fast and as long as possible. A harness supporting part of their body weight is used if needed. Assistance from a trainer is used if needed. A physical therapist supervises the training. Training is 5x/wk for 2 months, followed by a 2-month rest period. Participants then returned for Precision Training 5x/wk for 2 months. Participants train to walk over ground on 15 m straight hallway with obstacles they must step over, and targets they must step onto. This is followed by another 2-month rest.
- Precision First: Participants start with Precision Training. Participants train to walk over ground on 15 m straight hallway with obstacles they must step over, and targets they must step onto. Training is 5x/wk for 2 months, followed by a 2-month rest period. Participants then returned for Endurance Training 5x/wk for 2 months. Participants are trained to walk on a treadmill for as fast and as long as possible. A harness supporting part of their body weight is used if needed. Assistance from a trainer is used if needed. A physical therapist supervises the training, which is followed by another 2-month rest.
Period: Training Phase 1
Arm/Group | Endurance First | Precision First
Started | 10 | 11
Completed | 9 | 10
Not Completed | 1 | 1
Not completed — Format of intervention differed | 1 | 0
Not completed — Poor participation in intervention | 0 | 1
Period: Rest Phase 1
Arm/Group | Endurance First | Precision First
Started | 9 | 10
Completed | 9 | 9
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Training Phase 2
Arm/Group | Endurance First | Precision First
Started | 10 (1st subject didn't use same training(phase 1) as subsequent participants Phase 1 and 2 data removed.) | 9
Completed | 10 | 8
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Rest Phase 2
Arm/Group | Endurance First | Precision First
Started | 10 | 8
Completed | 8 | 7
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Endurance First: Participants start with Endurance Training. Participants are trained daily to walk on a treadmill for as fast and as long as possible. A harness supporting part of their body weight is used if needed. Assistance from a trainer is used if needed. A physical therapist supervises the training. Training is 5x/wk for 2 months, followed by a 2-month rest period. Participants then returned for training in the Precision Training 5x/wk for 2 months.Participants train to walk over ground on 15 m straight hallway with obstacles they must step over, and targets they must step onto. This is followed by another 2-month rest.
- Precision First: Participants start with Precision Training. Participants train to walk over ground on 15 m straight hallway with obstacles they must step over, and targets they must step onto. Training was 5x/wk for 2 months, followed by a 2-month rest period. Participants then returned for Endurance Training 5x/wk for 2 months. Participants are trained to walk on a treadmill for as fast and as long as possible. A harness supporting part of their body weight is used if needed. Assistance from a trainer is used if needed. A physical therapist supervises the training. followed by another 2-month rest.
- Total: Total of all reporting groups
Arm/Group | Endurance First | Precision First | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (14.4) | 44.0 (13.2) | 45.9 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Spinal Cord Injury - Functional Ambulation Profile (SCI-FAP) at Completion of Study
Description: This is a 7 item, timed walking test. Participants perform each of the walking tasks and the time to complete each task is recorded. Maximum times are set for each task. An assistance category is assigned based on the walking aids used, with 1 being no aid and 6 being unable to complete the task. A score for each item is calculated as: Time x Assistance factor/Mean able bodied time. A composite (single) score is obtained by summing the scores for all 7 items. The maximum score for the scale is 2100 indicating that the participant was unable to complete any of the 7 tasks within the allowed time. A minimum score of 7 indicates that all tasks were performed with no aids and at the mean able-bodied time. Results are reported as a measure of change: Final score - initial score. A negative result indicates improvement.
Time Frame: Change from Baseline I to the end of the study (i.e., end of Rest Period II, which was ~8 months after the beginning of the study)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Endurance First: Participants start with Endurance Training. Participants are trained daily to walk on a treadmill as fast and as long as possible. A harness supporting part of their body weight is used if needed. Assistance from a trainer is used if needed. A physical therapist supervises the training. Training is 5x/wk for 2 months, followed by a 2-month rest period. Participants then return for the Precision Training 5x/wk for 2 months.Participants train to walk over ground on 15 m straight hallway with obstacles they must step over, and targets they must step onto. This is followed by another 2-month rest.
- Precision First: Participants start with Precision Training. Participants train to walk over ground on 15 m straight hallway with obstacles they must step over, and targets they must step onto. Training is 5x/wk for 2 months, followed by a 2-month rest period. Participants then return for Endurance Training 5x/wk for 2 months. Participants are trained to walk on a treadmill for as fast and as long as possible. A harness supporting part of their body weight is used if needed. Assistance from a trainer is used if needed. A physical therapist supervises the training. followed by another 2-month rest.
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 8 | 8
units on a scale | -128.77 (180.73) | -64.07 (77.24)

2. Secondary Outcome: Change in Spinal Cord Injury - Functional Ambulation Profile (SCI-FAP) at 2 Months of Training Phase I
Description: as for outcome 1
Time Frame: Change from Baseline I to 2 months of Training Phase I
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Endurance First: Participants start with Endurance Training. Participants are trained daily to walk on a treadmill for as fast and as long as possible. A harness supporting part of their body weight is used if needed. Assistance from a trainer is used if needed. A physical therapist supervises the training. Trainingis 5x/wk for 2 months, followed by a 2-month rest period. Participants then return for training in the Precision Training 5x/wk for 2 months.Participants train to walk over ground on 15 m straight hallway with obstacles they must step over, and targets they must step onto. This is followed by another 2-month rest.
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 10
units on a scale | -129.09 (165.06) | -69.51 (106.51)

3. Secondary Outcome: Change in Spinal Cord Injury - Functional Ambulation Profile (SCI-FAP) at the End of 2 Months of Rest Period I
Description: as for outcome 1
Time Frame: Change from the end of Phase I training (measured at 2 months of Training Phase I) to 2 months of Rest Period I
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Endurance First: Participants start with Endurance Training. Participants are trained daily to walk on a treadmill for as fast and as long as possible. A harness supporting part of their body weight is used if needed. Assistance from a trainer is used if needed. A physical therapist supervises the training. Training is 5x/wk for 2 months, followed by a 2-month rest period. Participants then return for training in the Precision Training 5x/wk for 2 months.Participants train to walk over ground on 15 m straight hallway with obstacles they must step over, and targets they must step onto. This is followed by another 2-month rest.
- Precision First: Participants start with Precision Training. Participants train to walk over ground on 15 m straight hallway with obstacles they must step over, and targets they must step onto. Training is 5x/wk for 2 months, followed by a 2-month rest period. Participants then return for Endurance Training 5x/wk for 2 months. Participants are trained to walk on a treadmill for as fast and as long as possible. A harness supporting part of their body weight is used if needed. Assistance from a trainer is used if needed. A physical therapist supervises the training. This is followed by another 2-month rest.
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 9
units on a scale | -1.04 (49.67) | 10.34 (74.23)

4. Secondary Outcome: Change in Spinal Cord Injury - Functional Ambulation Profile (SCI-FAP) at 2 Months of Training Phase II
Description: as for outcome 1
Time Frame: Change from Baseline II to 2 months of Training Phase II
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 10 | 8
units on a scale | -15.28 (31.74) | -13.35 (31.58)
Statistical Analysis 1: Comparison: Endurance First; Test type: Superiority or Other; p = 0.04366667, t-test, 2 sided

5. Secondary Outcome: Change in Spinal Cord Injury - Functional Ambulation Profile (SCI-FAP) at the End of 2 Months of Rest Period II
Description: as for outcome 1
Time Frame: Change from the end of Phase II training (measured at 2 months of Training Phase II) to 2 months of Rest Period II
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 8 | 8
units on a scale | 1.61 (34.13) | 16.10 (63.86)

6. Secondary Outcome: Change in 6 Minute Walk Test (6MWT) at 2 Months of Training Phase I
Description: Participants walk for as far as possible in 6 min along a 25m hallway.
Time Frame: Change from Baseline I to 2 months of Training Phase I
Measure: Mean (Standard Deviation); unit: metres
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 10
metres | 32.75 (40.07) | 17.43 (26.67)

7. Secondary Outcome: Change in 6 Minute Walk Test (6MWT) at the End of 2 Months of Rest Period I
Description: Participants walk for as far as possible in 6 min along a 25m hallway. Total distance walked in the time is measured. Results are calculated as : Distance walked at end of period - Distance walked at beginning of period.
Time Frame: Change from the end of Phase I training (measured at 2 months of Training Phase I) to 2 months of Rest Period I
Measure: Mean (Standard Deviation); unit: metres
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 9
metres | 6.78 (32.69) | 32.23 (46.41)

8. Secondary Outcome: Change in 6 Minute Walk Test (6MWT) at 2 Months of Training Phase II
Description: as for outcome 7
Time Frame: Change from Baseline II to 2 months of Training Phase II
Measure: Mean (Standard Deviation); unit: metres
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 10 | 8
metres | 3.9 (11.11) | 25.78 (26.60)

9. Secondary Outcome: Change in 6 Minute Walk Test (6MWT) at the End of 2 Months of Rest Period II
Description: as for outcome 7
Time Frame: Change from the end of Phase II training to 2 months of Rest Period II
Measure: Mean (Standard Deviation); unit: metres
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 8 | 8
metres | -14.63 (29.94) | 17.00 (23.60)

10. Secondary Outcome: Change in 10 Metre Walk Test at a Self-selected Speed [10MWT(ss)] at 2 Months of Training Phase I
Description: Participants walk along a 14 meter path on a smooth floor at a comfortable pace. The middle 10 m is timed. Speed over 10 m is calculated as 10 m/Time. Results are calculated as: Final speed - initial speed.
Time Frame: Change from Baseline I to 2 months of Training Phase I
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 10
m/s | 0.07 (0.06) | 0.06 (0.08)

11. Secondary Outcome: Change in 10 Meter Walk Test at a Self-selected Speed [10MWT(ss)] at the End of 2 Months of Rest Period I
Description: as for outcome 10
Time Frame: Change from the end of Phase I training (measured at 2 months of Training Phase I) to 2 months of Rest Period I
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 9
m/s | 0.04 (0.12) | 0.09 (0.19)

12. Secondary Outcome: Change in 10 Meter Walk Test at a Self-selected Speed [10MWT(ss)] at 2 Months of Training Phase II
Description: as for outcome 10
Time Frame: Change from Baseline II to 2 months of Training Phase II
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 10 | 8
m/s | 0.02 (0.04) | 0.06 (0.15)

13. Secondary Outcome: Change in 10 Meter Walk Test at a Self-selected Speed [10MWT(ss)] at the End of 2 Months of Rest Period II
Description: as for outcome 10
Time Frame: Change from the end of Phase II training (measured at 2 months of Training Phase II) to 2 months of Rest Period II
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 8 | 8
m/s | -0.02 (0.12) | -0.09 (0.30)

14. Secondary Outcome: Change in 10 Meter Walk Test at a Fast Speed [10MWT(f)] at 2 Months of Training Phase I
Description: Participants walk as quickly as they are able to along a 14 meter path on a smooth floor. The middle 10 m is timed. Speed over 10 m is calculated as 10 m/Time. Results are calculated as: Final speed - initial speed.
Time Frame: Change from Baseline I to 2 months of Training Phase I
Population: Measure was added to study protocol midway through study. 5 out of 19 participants did not complete this measure at this time point. Data analysed for all participants who performed this measure.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 8 | 6
m/s | 0.07 (0.09) | 0.21 (0.20)

15. Secondary Outcome: Change in 10 Meter Walk Test at a Fast Speed [10MWT(f)] at the End of 2 Months of Rest Period I
Description: as for outcome 14
Time Frame: Change from the end of Phase I training (measured at 2 months of Training Phase I) to 2 months of Rest Period I
Population: Measure was added to study protocol midway through study. 4 out of 18 participants did not complete this measure at this time point. Data analysed for all participants who performed this measure.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 5
m/s | 0.04 (0.18) | 0.14 (0.11)

16. Secondary Outcome: Change in 10 Meter Walk Test at a Fast Speed [10MWT(f)] at 2 Months of Training Phase II
Description: as for outcome 14
Time Frame: Change from Baseline II to 2 months of Training Phase II
Population: Measure was added to study protocol midway through study. 3 out of 18 participants did not complete this measure at this time point. Data analysed for all participants who performed this measure.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 6
m/s | 0.06 (0.09) | 0.09 (0.13)

17. Secondary Outcome: Change in 10 Meter Walk Test at a Fast Speed [10MWT(f)] at the End of 2 Months of Rest Period II
Description: as for outcome 14
Time Frame: Change from the end of Phase II training (measured at 2 months of Training Phase II) to 2 months of Rest Period II
Population: Measure was added to study protocol midway through study. 2 out of 16 participants did not complete this measure at this time point. Data analysed for all participants who performed this measure.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 7 | 7
m/s | -0.09 (0.11) | 0.12 (0.28)

18. Secondary Outcome: Change in Walking Index for Spinal Cord Injury Version II Self-selected (WISCI-II ss) at 2 Months of Training Phase I
Description: Participants are scored from 0 to 20 based on the walking aid they select to walk a distance of 10 meters. Walking aids and physical assistance provided are ranked on an ordinal scale from 1 to 20. A score of 0 indicates the participant is unable to walk 10 m, 20 indicates no aids are required to complete the task.
  Results are reported as Final score - Initial score. A positive result indicates that less assistance was required.
Time Frame: Change from Baseline I to 2 months of Training Phase I
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 10
units on a scale | 0.32 (0.65) | 1.30 (2.21)

19. Secondary Outcome: Change in Walking Index for Spinal Cord Injury Version II Self-selected (WISCI-II ss) at the End of 2 Months of Rest Period I
Description: as for outcome 18
Time Frame: Change from the end of Phase I training (measured at 2 months of Training Phase I) to 2 months of Rest Period I
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 9
units on a scale | -0.22 (0.67) | -0.22 (1.09)

20. Secondary Outcome: Change in Walking Index for Spinal Cord Injury Version II Self-selected (WISCI-II ss) at 2 Months of Training Phase II
Description: as for outcome 18
Time Frame: Change from Baseline II to 2 months of Training Phase II
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 10 | 8
units on a scale | 0.50 (1.58) | 0 (0)

21. Secondary Outcome: Change in Walking Index for Spinal Cord Injury Version II Self-selected (WISCI-II ss) at the End of 2 Months of Rest Period II
Description: as for outcome 18
Time Frame: Change from the end of Phase II training (measured at 2 months of Training Phase II) to 2 months of Rest Period II
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 8 | 8
units on a scale | 0 (0) | 0 (0)

22. Secondary Outcome: Change in Walking Index for Spinal Cord Injury Version II Maximum [WISCI-II (Max)] at 2 Months of Training Phase I
Description: Participants are scored from 0 to 20 based on the least amount of assistance/aid they require to walk a distance of 10 meters. Walking aids and physical assistance provided are ranked on an ordinal scale from 1 to 20. A score of 0 indicates the participant is unable to walk 10 m, 20 indicates no aids are required to complete the task.
  Results are reported as Final score - Initial score. A positive result indicates that less assistance was required.
Time Frame: Change from Baseline I to 2 months of Training Phase I
Population: Measure was added to study protocol midway through study. 3 out of 19 participants did not complete this measure at this time point. Data analysed for all participants who performed this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 8 | 8
units on a scale | 0.73 (1.08) | 1.63 (2.39)

23. Secondary Outcome: Change in Walking Index for Spinal Cord Injury Version II Maximum [WISCI-II (Max)] at the End of 2 Months of Rest Period I
Description: as for outcome 22
Time Frame: Change from the end of Phase I training (measured at 2 months of Training Phase I) to 2 months of Rest Period I
Population: Measure was added to study protocol midway through study. 2 out of 17 participants did not complete this measure at this time point. Data analysed for all participants who performed this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 8 | 8
units on a scale | -0.25 (0.53) | -0.19 (0.75)

24. Secondary Outcome: Change in Walking Index for Spinal Cord Injury Version II Maximum [WISCI-II (Max)] at 2 Months of Training Phase II
Description: as for outcome 22
Time Frame: Change from Baseline II to 2 months of Training Phase II
Population: Measure was added to study protocol midway through study. 1 out of 18 participants did not complete this measure at this time point. Data analysed for all participants who performed this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 8
units on a scale | 0.22 (1.33) | 0.44 (1.59)

25. Secondary Outcome: Change in Walking Index for Spinal Cord Injury Version II Maximum [WISCI-II (Max)] at the End of 2 Months of Rest Period II
Description: as for outcome 22
Time Frame: Change from the end of Phase II training (measured at 2 months of Training Phase II) to 2 months of Rest Period II
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 8 | 8
units on a scale | 0.00 (0.00) | -0.50 (1.41)

26. Secondary Outcome: Change in Activities-specific Balance Confidence Scale (ABC) at 2 Months of Training Phase I
Description: A survey with 16 questions regarding the participants confidence in their ability to perform specific tasks requiring balance. Participants rate their confidence as a percentage from 0% (no confidence in their ability to perform the task) to 100% 9 completely confident in their ability to complete the task safely. Total score is calculated as: Sum of item scores/16 and is expressed as a percentage.
  Results are reported as Final score - Initial score. A positive result indicates a higher level of confidence in ability.
Time Frame: Change from Baseline I to 2 months of Training Phase I
Measure: Mean (Standard Deviation); unit: percentage of confidence in balance
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 10
percentage of confidence in balance | 4.15 (9.54) | 3.15 (8.79)

27. Secondary Outcome: Change in Activities-specific Balance Confidence Scale (ABC) at the End of 2 Months of Rest Period I
Description: as for outcome 26
Time Frame: Change from the end of Phase I training (measured at 2 months of Training Phase I) to 2 months of Rest Period I
Measure: Mean (Standard Deviation); unit: percentage of confidence in balance
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 9
percentage of confidence in balance | 0.38 (8.23) | 1.70 (3.90)

28. Secondary Outcome: Change in Activities-specific Balance Confidence Scale (ABC) at 2 Months of Training Phase II
Description: as for outcome 26
Time Frame: Change from Baseline II to 2 months of Training Phase II
Measure: Mean (Standard Deviation); unit: Percentage of confidence in balance
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 10 | 8
Percentage of confidence in balance | 3.78 (5.37) | 6.48 (10.52)

29. Secondary Outcome: Change in Activities-specific Balance Confidence Scale (ABC) at the End of 2 Months of Rest Period II
Description: as for outcome 26
Time Frame: Change from the end of Phase II training (measured at 2 months of Training Phase II) to 2 months of Rest Period II
Measure: Mean (Standard Deviation); unit: percentage of confidence in balance
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 8 | 8
percentage of confidence in balance | -0.08 (5.20) | -0.63 (5.44)

30. Secondary Outcome: Change in Center for Epidemiologic Studies - Depression Scale (CES-D) at 2 Months of Training Phase I
Description: A 20 question survey to measure current level of depressive symptoms. The participant ranks their emotional state or actions for each question on an ordinal scale of 0 to 3, with 0 indicating rarely or never and 3 being most of the time. A minimum score of 0 indicates no depressive symptoms, and a score of 10 or greater is considered indicative of depression. The max score for the scale is 60.
  Results are reported as Final score - Initial score. A negative result indicates a lower level of depression.
Time Frame: Change from Baseline I to 2 months of Training Phase I
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 10
units on a scale | -3.85 (5.40) | -2.42 (6.95)

31. Secondary Outcome: Change in Center for Epidemiologic Studies - Depression Scale (CES-D) at the End of 2 Months of Rest Period I
Description: A 20 question survey to measure current level of depressive symptoms.The participant ranks their emotional state or actions for each question on an ordinal scale of 0 to 3, with 0 indicating rarely or never and 3 being most of the time. A minimum score of 0 indicates no depressive symptoms, and a score of 10 or greater is considered indicative of depression. The max score for the scale is 60.
  Results are reported as Final score - Initial score. A negative result indicates a lower level of depression.
Time Frame: Change from the end of Phase I training (measured at 2 months of Training Phase I) to 2 months of Rest Period I
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 9
units on a scale | 0.61 (1.98) | -0.64 (3.27)

32. Secondary Outcome: Change in Center for Epidemiologic Studies - Depression Scale (CES-D) at 2 Months of Training Phase II
Description: as for outcome 31
Time Frame: Change from Baseline II to 2 months of Training Phase II
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 10 | 8
units on a scale | -2.75 (2.95) | -0.53 (3.70)

33. Secondary Outcome: Change in Center for Epidemiologic Studies - Depression Scale (CES-D) at the End of 2 Months of Rest Period II
Description: as for outcome 31
Time Frame: Change from the end of Phase II training (measured at 2 months of Training Phase II) to 2 months of Rest Period II
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 8 | 8
units on a scale | 3.25 (5.92) | -0.25 (3.24)

34. Secondary Outcome: Change in Manual Muscle Test (MMT) at 2 Months of Training Phase I
Description: The strength of each of 8 major muscle groups (per side) in the lower extremities is graded using the standard manual muscle testing technique. Strength is graded from 0 (no muscle activity detected) to 5 (strength with normal range for the muscle group). Scores from all muscle groups are added to obtain the total score. The total score ranges from 0 (unable to produce any muscle activity in all 8 muscle groups bilaterally) to 80 (normal strength in all 8 muscle groups bilaterally).
  Results are reported as Final score - Initial score. A positive result indicates an increase in strength.
Time Frame: Change from Baseline I to 2 months of Training Phase I
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 10
units on a scale | 1.29 (2.51) | 2.50 (5.60)

35. Secondary Outcome: Change in Manual Muscle Test (MMT) at the End of 2 Months of Rest Period I
Description: as for outcome 34
Time Frame: Change from the end of Phase I training (measured at 2 months of Training Phase I) to 2 months of Rest Period I
Population: This measure was accidentally omitted for 1 participant at the end of this phase. Data analysed for all participants who performed this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 8 | 8
units on a scale | -2.45 (4.19) | -1.06 (3.13)

36. Secondary Outcome: Change in Manual Muscle Test (MMT) at 2 Months of Training Phase II
Description: as for outcome 34
Time Frame: Change from Baseline II to 2 months of Training Phase II
Population: This measure was accidentally omitted for 1 participant at beginning of this phase. Data analysed for all participants who performed this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 8
units on a scale | 1.22 (2.90) | 0.56 (3.21)

37. Secondary Outcome: Change in Manual Muscle Test (MMT) at the End of 2 Months of Rest Period II
Description: as for outcome 34
Time Frame: Change from the end of Phase II training (measured at 2 months of Training Phase II) to 2 months of Rest Period II
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 8 | 8
units on a scale | -3.00 (3.36) | 0.07 (4.76)

38. Secondary Outcome: Change in Cutaneomuscular Reflexes at 2 Months of Training Phase I
Description: Reflexes are elicited in standing by electrical stimulation (3 pulses) of the tibial nerve at the ankle using surface electrodes. Responses are recorded with surface electromyography (EMG) in µV.
Time Frame: Change from Baseline I to 2 months of Training Phase I
Population: Data from 6 participants could not be analysed due to absence of reflex, or difficulty with EMG signals. Remaining 13 were analysed.
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 6 | 7
µV | -6.84 (6.00) | 2.36 (17.35)

39. Secondary Outcome: Change in Cutaneomuscular Reflexes at the End of 2 Months of Rest Period I
Description: Reflexes are elicited with electrical stimulation (3 pulses) of the tibial nerve at the ankle using surface electrodes. Responses are recorded with surface electromyography (EMG). Responses are typically recorded in standing.
Time Frame: Change from the end of Phase I training (measured at 2 months of Training Phase I) to 2 months of Rest Period I
Population: Data was analysed for the 13 participants who provided CMR data in Training phase 1 in order to dtermine if training effect was maintained. 1 out 13 withdrew and 1 did not produce adequate reflex activity to allow analysis
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 5 | 6
µV | 0.18 (5.60) | 4.35 (6.92)

40. Secondary Outcome: Change in Cutaneomuscular Reflexes at 2 Months of Training Phase II
Description: as for outcome 39
Time Frame: Change from Baseline II to 2 months of Training Phase II
Population: Data from 5 participants could not be analysed due to absence of reflex, or difficulty with EMG signals. Remaining 13 were analysed.
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 7 | 6
µV | 3.01 (7.09) | -5.97 (11.14)

41. Secondary Outcome: Change in Cutaneomuscular Reflexes at the End of 2 Months of Rest Period II
Description: as for outcome 39
Time Frame: Change from the end of Phase II training (measured at 2 months of Training Phase II) to 2 months of Rest Period II
Population: Data was analysed for the 13 participants who provided CMR data in Training phase 1 to determine whether training effect was maintained. 1 out 13 withdrew and 3 did not produce adequate reflex activity to allow analysis.
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 4 | 5
µV | 2.13 (5.56) | 1.82 (14.42)

42. Secondary Outcome: Change in Transcranial Magnetic Stimulation (TMS) at 2 Months of Training Phase I
Description: Single-pulse TMS is applied over the motor cortex, and electromyographic responses are recorded in the tibialis anterior muscles on both legs.
Time Frame: Change from Baseline I to 2 months of Training Phase I
Measure: Mean (Standard Error); unit: Percentage of baseline mep
Groups:
- Precision First: Participants start with Precision Training. Participants train to walk over ground on 15 m straight hallway with obstacles they must step over, and targets they must step onto. Training is 5x/wk for 2 months, followed by a 2-month rest period. Participants then return for Endurance Training 5x/wk for 2 months. Participants are trained to walk on a treadmill for as fast and as long as possible. A harness supporting part of their body weight can be used if needed. Assistance from a trainer is used if needed. A physical therapist supervises the training. This is followed by another 2-month rest.
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 7
Percentage of baseline mep | 122.9 (7.8) | 113.9 (9.0)

43. Secondary Outcome: Change in Transcranial Magnetic Stimulation (TMS) at the End of 2 Months of Rest Period I
Description: as for outcome 42
Time Frame: Change from the end of Phase I training (measured at 2 months of Training Phase I) to 2 months of Rest Period I
Measure: Mean (Standard Error); unit: percentage of baseline mep
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 7
percentage of baseline mep | 115.1 (14.2) | 121.7 (7.1)

44. Secondary Outcome: Change in Transcranial Magnetic Stimulation (TMS) at 2 Months of Training Phase II
Description: as for outcome 42
Time Frame: Change from Baseline II to 2 months of Training Phase II
Measure: Mean (Standard Error); unit: percentage of baseline mep
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 9 | 7
percentage of baseline mep | 124.3 (12.4) | 111.0 (9.7)

45. Secondary Outcome: Change in Transcranial Magnetic Stimulation (TMS) at the End of 2 Months of Rest Period II
Description: Maximum evoked potentials were measured and compared to baseline measures for major muscle groups.
Time Frame: Change from the end of Phase II training (measured at 2 months of Training Phase II) to 2 months of Rest Period II
Measure: Mean (Standard Error); unit: percentage of baseline MEP
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 7 | 6
percentage of baseline MEP | 141.0 (17.1) | 111.6 (10.4)

46. Secondary Outcome: Change in Electromyography During Treadmill Walking at 2 Months of Training Phase I
Description: Participants walk on a treadmill at a variety of speeds while we record surface electromyography from leg muscles and motion data from electrogoniometers place on the knees.
Time Frame: Change from Baseline I to 2 months of Training Phase I
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 6 | 7
µV | 0.28 (3.76) | 0.14 (5.24)

47. Secondary Outcome: Change in Electromyography During Treadmill Walking at the End of 2 Months of Rest Period I
Description: as for outcome 46
Time Frame: Change from the end of Phase I training (measured at 2 months of Training Phase I) to 2 months of Rest Period I
Population: Data was analysed for the 13 participants who provided CMR data in Training phase 1 to determine if training effect was maintained. 1 out 13 withdrew and 1 did not produce adequate reflex activity to allow analysis
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 5 | 6
µV | 1.04 (3.54) | 0.38 (6.43)

48. Secondary Outcome: Change in Electromyography During Treadmill Walking at 2 Months of Training Phase II
Description: as for outcome 46
Time Frame: Change from Baseline II to 2 months of Training Phase II
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 7 | 6
µV | 0.73 (2.76) | -0.26 (7.73)

49. Secondary Outcome: Change in Electromyography During Treadmill Walking at the End of 2 Months of Rest Period II
Description: as for outcome 46
Time Frame: Change from the end of Phase II training (measured at 2 months of Training Phase II) to 2 months of Rest Period II
Population: Data was analysed for the 13 participants who provided CMR data in Training phase 1. 1 out 13 withdrew and 3 did not produce adequate reflex activity to allow analysis.
Measure: Mean (Standard Deviation); unit: µV
Arm/Group | Endurance First | Precision First
Number analyzed (Participants) | 4 | 5
µV | 0.53 (3.11) | 0.63 (6.17)

ADVERSE EVENTS:
Arm/Group | Endurance First | Precision First
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

LIMITATIONS AND CAVEATS:
* Participants were a sample of convenience, likely the most highly motivated due to the time commitment.
* Sample size was small.
* 4 participants were less than 1 year post injury and may have had spontaneous recovery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No